CLINICAL TRIAL: NCT04508491
Title: The Best Treatment Strategy for the Reservation of Cognitive Function in Patients With Persisted Atrial Fibrillation
Brief Title: Cognitive Function in Patients With Persisted Atrial Fibrillation
Acronym: SMART-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201912175RINC
Record Dates: First submitted 2020-08-09; First posted 2020-08-11 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation, Persistent; Cognitive Function
Keywords: Atrial Fibrillation; Cognitive Function
MeSH Terms: conditions — Atrial Fibrillation | interventions — Heart Rate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythm control (Experimental): Rhythm control with medication or any procedure
  Interventions: Other: Rhythm control
- Rate control (Active Comparator): Rate control with medication or any procedure
  Interventions: Other: Rate control

INTERVENTIONS:
Other: Rhythm control — Rhythm control with medications or any procedure
  Arms: Rhythm control
Other: Rate control — Rate control
  Arms: Rate control

SUMMARY:
Compare the difference of cognitive function between different treatment strategy in patients with persistent atrial fibrillation

DETAILED DESCRIPTION:
The prevalence of atrial fibrillation (AF) had been increasing for the past decade. The increase of AF was attributed to the aging of the population and the increased awareness of the disease among people and the primary physicians. However, we have not achieved the consensus whether aggressive rhythm control or conservative rate control is better in a patient with asymptomatic persisted AF. We do prescribe anti-coagulant for stroke prevention, but which treatment strategy is best for the patients is uncertain.

The clinical trial of catheter-based ablation for rhythm control compared to traditional medication control has not shown the benefit of reducing all-cause mortality, but it did show a reduction of re-hospitalization and the recurrence of AF. On the contrary, the study in heart failure patients had shown a significant benefit applying catheter-based rhythm control strategy to reduce all-cause mortality. The different results of these two trials told us the benefit of rhythm control is not easily to be seen in a short-term, but could be seen in a long term or in high risk patients. The association between AF and cognitive impairment has also been reported in observation cohort. However, there is no sold evidence in clinical trials to show the improvement of cognitive function by treating atrial fibrillation. One study did show improvement of cognitive function with questionnaire, but the other showed new lesion detected by traditional magnetic resonance imaging (MRI) after ablation, though the lesion resolved after one year of follow-up. There is no clear answer to which treatment strategy is better for the patients' cognitive function。 Therefore, we designe a prospective, randomized, blind endpointtrial. We will enroll the patients with persisted AF, and use advanced MRI (DTI/SWI) and questionnaire to longitudinally study the cognitive function change of the patients before and after the initiation of anti-coagulant agents, before and after the catheter-based ablation, and use this as a surrogate to understand the best treatment strategy for these AF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Those who meet the diagnosis of persistent atrial fibrillation, meet one of the following conditions:

   * The twelve-lead electrocardiogram is used to diagnose atrial fibrillation, and to cooperate with clinical diagnosis.
   * 24 hours ECG diagnosis 100% atrial fibrillation, with clinical diagnosis.
   * The seven-day ECG recorder diagnosed 100% atrial fibrillation.
2. Willing to accept treatment recommended by doctors, containing anticoagulant, and cooperate with examination and treatment in the coming year.

Exclusion Criteria:

1. Unwilling to sign the clinical trial consent form.
2. Unable to complete the cognitive function questionnaire.
3. Unable to complete brain MRI examination due to various reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2025-02-26 (Actual)

PRIMARY OUTCOMES:
Cognitive function | 12 months
  MOCA questionnaire
Cognitive function | 12 months
  brain MRI

SECONDARY OUTCOMES:
Quality of Life questionnaire | 12 months
  SF-36 questionnaire
Hospitalization for cardiovascular cause | 12 months
all cause mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No